CLINICAL TRIAL: NCT05184920
Title: CSD201004: An Actual Use Study of P10 and P13 Nicotine Pouches Among U.S. Adult Smokers
Status: Completed | Type: Observational
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CSD201004
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Smoking; Tobacco Use; Tobacco Smoking
MeSH Terms: conditions — Smoking; Tobacco Use; Tobacco Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: P1012919 nicotine pouch — P1012919, a nicotine pouch with 12 mg of nicotine
Other: P1012915 nicotine pouch — P1012915, a nicotine pouch with 8 mg of nicotine
Other: P1012914 nicotine pouch — P1012914, a nicotine pouch with 4 mg of nicotine
Other: P1013315 nicotine pouch — P1013315, a nicotine pouch with 8 mg of nicotine
Other: P1013119 nicotine pouch — P1013119, a nicotine pouch with 12 mg of nicotine
Other: P1013218 nicotine pouch — P1013218, a nicotine pouch with 10 mg of nicotine
Other: P1012818 nicotine pouch — P1012818, a nicotine pouch with 10 mg of nicotine
Other: P1312915 nicotine pouch — P1312915, a nicotine pouch with 8 mg of nicotine
Other: P1312914 nicotine pouch — P1312914, a nicotine pouch with 4 mg of nicotine
Other: P1313015 nicotine pouch — P1313015, a nicotine pouch with 8 mg of nicotine
Other: P1313314 nicotine pouch — P1313314, a nicotine pouch with 4 mg of nicotine
Other: P1312815 nicotine pouch — P1312815, a nicotine pouch with 8 mg of nicotine

SUMMARY:
The purpose of this Actual Use Study (AUS) is to investigate how U.S. adult tobacco consumers 21-60 years of age) who are regular smokers (≥5 cigarettes/day) on at least 20 days out of the past 30 days will use P10 and P13 nicotine pouches (Study Investigational Product [IP]) over a 6-week Actual Use Period (AUP) in their real-life/naturalistic environment and in the context of typical consumer marketing materials. Subjects will self-report their ad libitum use of the Study IP as well as use of combustible cigarette (CC) and any other tobacco- or nicotine-containing product (TNP) on a daily basis using an electronic diary (eDiary). The study design is planned to address topics that FDA's Center for Tobacco Products (CTP) has identified as useful in evaluating new tobacco products.

DETAILED DESCRIPTION:
The AUS is a multi-site, open-label, 8-week, prospective observational study, conducted at multiple sites geographically dispersed within the U.S.

Adult smokers will be recruited, and candidate subjects who meet study inclusion criteria and none of the exclusion criteria will give verbal consent for further screening. Candidate subjects will be scheduled to attend an in-person Site Enrollment Visit (SEV).

At the SEV, site staff will confirm eligibility, including age verification with a government-issued photo identification. Candidate subjects will review product information and will be shown physical examples of the Study IP, but will not sample the products. Those who indicate an "intention to use" the Study IP will undergo a second consent process, will be enrolled in the study, and will install and be trained on an eDiary application on their personal smartphones or site provisioned devices.

During a 1-week Baseline Assessment Period (BAP, Week 0), enrolled subjects will record all CC and any other TNP use in the eDiary. At the end of the BAP, subjects will return to the study site for Site Visit 1 (SV1). At this visit, subjects will be able to select up to five different Study IPs for the first two weeks of the AUP from the Study IPs available.

During the subsequent 6-week observational AUP, subjects can choose to use the Study IP (or not). Subjects will be instructed to record all daily Study IP, TNP and CC use in the eDiary. They will return to the site every two weeks during the AUP for an in-person interview to answer questionnaires and for product accountability and resupply. As with SV1, at Site Visit 2 (SV2) and Site Visit 3 (SV3), subjects will be able to select up to five IP varieties (if desired) for use during the subsequent 2-week AUP. After Week 6 of the AUP, there will be a final site visit (SV4) and week-long Close Out Period (COP).

In addition to collecting information on daily ad libitum use of Study IP, TNP and CC use, the study will assess subjective measures (i.e., product assessment) for each Study IP, including product use behaviors and intent to use again (at close of study). Information on intention to quit CC will be collected at enrollment and at study conclusion. A passive surveillance mechanism will be used to collect information on adverse health experiences.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or females, 21-60 years old, inclusive, verified with government-issued photo ID.
2. Must be a current smoker of factory-made filtered menthol and/or non-menthol cigarettes, has smoked at least 100 cigarettes in their lifetime, and typically smokes on at least 20 days out of the past 30 days.
3. Smokes on average ≥ 5 combustible cigarettes per day (CPD) on days when cigarettes are smoked. (There are no other requirements or exclusions regarding other TNP use. Dual and poly-users may enroll if they fulfill the cigarette use requirements.)
4. Must indicate "an intention to use" Study IP after a brief review of product information and product demonstration at the SEV. Subjects will not try the product at the SEV.
5. Available and interested in participating in an 8-week study about the Study IP.
6. Able and willing to comply with all study requirements, including questionnaires, the eDiary reporting procedures, and provide valid contact information.
7. Able to read, understand, and willing to sign Informed Consent Forms (ICFs) and complete questionnaires written in English.
8. Has not participated in any tobacco-, vapor-, or nicotine-related research within 3 months of screening.
9. Agrees that the IP received are for their own personal use and they will not share the product with others.
10. Agrees to restrict use of Study IP to only the investigational products (specified flavors, nicotine levels, and pouch sizes) supplied by the study Sponsor free of charge and labeled as "For Investigational Use Only" and to not obtain/use any other nicotine pouch products from other commercial sources.

Exclusion Criteria:

1. Self-reports as currently quitting or intending to quit within the next 3 months all tobacco or nicotine product use ("currently" is defined as within (≤) 30 days). Those who intend to quit CC only can be enrolled.
2. Must not be an ever-user of any nicotine pouches prior to screening.
3. Female subjects who are currently pregnant or breastfeeding or planning to become pregnant or start breastfeeding within the next 6 months based on self-report.
4. Female subjects who self-report they are not using adequate methods to prevent pregnancy.
5. Self-reports "poor" physical health (based on the five-category Population Assessment of Tobacco and Health (PATH) questionnaire): "In general, how would you rate your physical health?" (Response choices: Excellent, Very Good, Good, Fair, Poor).
6. Self-reports "poor" mental health (based on the five-category PATH questionnaire): "In general, how would you rate your mental health?" (Response choices: Excellent, Very Good, Good, Fair, Poor).
7. Employees of tobacco or vapor companies.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study sample will comprise approximately 1,200 generally healthy, U.S. adult tobacco consumer 21 to 60 years of age, inclusive, who are regular smokers (≥5 cigarettes/day) on at least 20 of the past 30 days, who are not currently quitting all TNP use, and who have no intention of quitting all TNP use in the next three months (intention of quitting CC use only is allowable). A recruiting target for younger smokers (21-30 years old) of approximately 15% will be established 15% to ensure that they are sufficiently represented among the enrolled subjects.
Sampling Method: Non-Probability Sample
Enrollment: 1105 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Number and Proportion of Established Users | 6 weeks
  Number and proportion of subjects who meet the definition of "established users" of the Study IP
Number and Proportion of Established Users who reduce their CPD consumption | 8 weeks
  Number and proportion of subjects among "established users" who reduce their CPD consumption by at least 50%
Descriptive weekly average CPD consumption | 8 weeks
  Descriptive weekly average CPD consumption per subject among all subjects who complete the study, including both established and non-established users of the Study IP

CONTACTS AND LOCATIONS:
Overall Officials: Patrudu Makena, PhD, Study Director — RAIS
Locations (10):
- United States (10):
  - Schlesinger Phoenix, Phoenix, Arizona
  - Schlesinger Atlanta, Atlanta, Georgia
  - Schlesinger Chicago, Chicago, Illinois
  - Schlesinger Kansas City, Kansas City, Missouri
  - Schlesinger St. Louis, St Louis, Missouri
  - Schlesinger New Jersey, Iselin, New Jersey
  - Schlesinger Columbus, Columbus, Ohio
  - Schlesinger Philadelphia, Philadelphia, Pennsylvania
  - Schlesinger Dallas, Dallas, Texas
  - Schlesinger Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No